CLINICAL TRIAL: NCT04513782
Title: The Contributions of Age Related Changes in the Sound Localization Pathway to Central Hearing Loss
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-1213; R01DC017924 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Healthy Individuals; Hearing Loss, Central
MeSH Terms: conditions — Hearing Loss, Central

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Audiological Assessments — Participants will all undergo routine audiological assessments. The results from these assessments will be evaluated in order to advance understanding of central hearing loss.

SUMMARY:
Age-related hearing loss, presbycusis, affects up to 50% of American adults. There are two main causes for presbycusis: 1) Progressive death of hair cells in the inner ear, and 2) Central hearing loss, or the reduced ability to decipher the sound source of interest from other competing sounds in a multi-source complex environment. The first cause is better understood and treatment options, such as hearing aids and cochlear implants, are available. However, central hearing loss is not as well understood and there is not a treatment available at this time. This study aims to advance our understanding of central hearing loss by evaluating the abilities of younger and older listeners in two primary outcome measures: to 1) neurologically process sound stimuli and 2) focus on conversational speech in the presence of spatially-separated competing background noise. A test using Auditory Brainstem Responses (ABR) will be used to evaluate the brain's response to clicking sounds.

This study will assess all waveform data, but will focus particularly on wave III. Sentence in noise tests will be used to assess each subject's ability to process speech in noisy situations. Both the ABR and sentence in noise tests are non-invasive and are commonly used in audiology practices to diagnosis and treat a variety of audiological pathologies.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ranges

   a. 21 years (inclusive) and 89years (inclusive)
2. Subjects exhibiting no poorer than a mild hearing loss, defined as hearing thresholds no worse than 40dBHL at any test frequency 250-4000 Hz based on pure tone audiometry
3. Subjects scoring 26 or higher on a screening measure of cognitive status (Montreal Cognitive Screening Assessment; MoCA)

Exclusion Criteria:

1. Patients outside the age range of 21-89
2. Patients with an air-bone gap greater than 10dBHL at any frequency
3. Patients who are decisionally challenged and/or unable to complete speech perception testing. These patients are excluded based on the study requiring behavioral responses to some tests
4. Patients with little command of the English language who are unable to understand and repeat back simple everyday English sentences.
5. Illiterate patients
6. Patients with neurodegenerative diseases.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Speech in Noise Performance | through study completion, an average of 6 years
  Auditory perception task requiring participants to discriminate speech sound in quiet and in back ground noise. Takes about 90min.
Auditory Brainstem Response | through study completion, an average of 6 years
  Non-invasive auditory electrophysiological measure of brainstem electrical activity captured using electrodes placed on the scalp while sounds are played to one or both ears. Takes about 60min
Spatial Acuity | through study completion, an average of 6 years
  Auditory perception task requiring participants to judge the location of a sound. Takes about 90min

SECONDARY OUTCOMES:
Working Memory Assessment | through study completion, an average of 6 years
  Reading span test to understand working memory capacity. Takes about 20min
Electrocorticogram | through study completion, an average of 6 years
  Non-invasive auditory electrophysiological measure of brainstem electrical activity captured using electrodes placed on the scalp while sounds are played to one or both ears. Takes about 45min.
Subject Questionnaires | through study completion, an average of 6 years
  Questionnaires administered to subject to gather information on health and hearing history, noise exposure, everyday listening. Takes about 30min.
TFS-AF | through study completion, an average of 6 years
  Two-alternative forced choice auditory perception task requiring participants to determine which sound has been modified. Takes about 20min.
Spectrotemporal Modulation | through study completion, an average of 6 years
  Two-alternative forced choice auditory perception task requiring participants to determine which sound has been modified. Takes about 30min

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tollin, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No